CLINICAL TRIAL: NCT02767336
Title: Project Bloom Regulatory Clinical Evaluation - System Accuracy, User Performance, System Use, Instructions for Use and Marketing Claims Evaluation
Brief Title: Project BLOOM Regulatory Clinical Evaluation - System Accuracy, User Performance and System Use Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeScan (Industry)
Collaborators: Bio-Kinetic Europe, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 3141352 and 3141353
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood Glucose monitoring System (BGMS) (Experimental): Intervention: Blood Glucose monitoring System (BGMS) Results obtained from the BGMS for UP and SA are compared to a reference instrument (YSI)
  Interventions: Device: Blood Glucose Monitoring System.

INTERVENTIONS:
Device: Blood Glucose Monitoring System. — In vitro diagnostic medical device

SUMMARY:
Clinical Evaluation including System Accuracy, User Performance, System Use, Instructions for Use and Marketing Claims Evaluation.

ELIGIBILITY:
Summary of Inclusion Criteria:

* Able to voluntarily provide written informed consent to participate in the study.
* User Performance Accuracy Testing Only: Self-Monitoring - Subject is currently performing unassisted self-monitoring of blood glucose.
* For subjects participating in the In Vivo Glucose adjustment procedure age range is 18 - 45.

Summary of Exclusion Criteria:

* Female subjects who are pregnant or lactating.
* Subjects who, in the opinion of the Investigator, are unsuitable for participation in the study.
* User Performance Accuracy Testing Only -Prior involvement with the investigational BGMS being used in this study.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2016-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
User Performance (UP) evaluation measured by blood glucose level (mg/dl) of BGMS vs reference instrument. | Up to 1 hour
  UP evaluation of blood glucose monitoring systems compared to a reference instrument. Samples collected by subject and HCP ( Health Care Professional)
System Accuracy (SA) evaluation measured by blood glucose level(mg/dl) of BGMSs vs reference instrument. | Up to 1 hour
  Accuracy verification of blood glucose monitoring systems compared to a reference instrument. Samples collected by HCP only.
System Use Evaluation questionnaire. | Up to 15 minutes
  Assessment of how the patient uses the BGMS.
Instructions for Use Evaluation questionnaire. | Up to 6 days.
  Questionnaires to assess the effectiveness of the instructions for use.
Marketing Claims Evaluation questionnaire. | Up to 6 days.
  Assess Lay User Acceptance of the Bloom BGMS in support of marketing claims.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Stewart, Study Director — LifeScan Scotland Ltd
Locations (4):
- United Kingdom (4):
  - BioKinetic Europe Ltd, Belfast, Antrim
  - Diabetes Centre, Heartlands Hospital, Birmingham
  - NHS Lothian, Edinburgh
  - Highland Diabetes Institute, Inverness

IPD SHARING:
Plan to Share IPD: No